CLINICAL TRIAL: NCT04094714
Title: CHACO Study: Control of Arterial Hypertension in Colombian Patients
Acronym: CHACO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scandinavia Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: CHACO
Record Dates: First submitted 2019-09-13; First posted 2019-09-19 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiological study (cross-sectional study) in order to determine the patients who present an adequate control of the Blood Pressure (BP), in a population of Colombian patients diagnosed with Arterial Hypertension (AH) and who are under pharmacological treatment.

DETAILED DESCRIPTION:
OBJECTIVE: To determine the proportion of patients who present an adequate control of the Blood Pressure (BP), in a population of Colombian patients diagnosed with Arterial Hypertension (AH) and who are under pharmacological treatment.

MATERIALS AND METHODS: Epidemiological study (cross-sectional study), multicentre type, in patients older than 18 years with prior diagnosis of AH in Colombia. The blood pressure control will be evaluated as the main variable (only one single blood pressure check in the doctor's office). Other secondary variables to evaluate are: demographical analysis, type (s) of antihypertensive treatment (s) used in patients, level of BP control, adverse events associated with antihypertensive treatment, comorbidities and risk factors, adherence, perception about the possible benefits of the use of combined therapy in "mono-tablet" versus "multi-tablet". The analysis will be carried out from two perspectives: A first descriptive approach and a second analytical approach, with a level of significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Prior diagnosis of Arterial Hypertension (AH) ≥ 3 months before
* Patients who are under pharmacological treatment of AH ≥ 3 months before

Exclusion Criteria:

* The patient has rejected the participation in the study.
* Patients who, in the judgment of the Investigator, do not understand or are not willing to adequately answer the questions.
* Mental or psychiatric illness that, in the judgment of the investigator, does not allow adequate information to be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colombian patients
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Patients with adequate control of the Blood Pressure (BP) | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years.
  Proportion of patients who present an adequate control of the Blood Pressure (BP)

SECONDARY OUTCOMES:
Demographic analysis | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years.
  Characterization of patients
Treatment analysis | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years.
  Characterization of treatment (s) used
Personal history of diseases | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years.
  Evaluation of personal history of diseases
Adverse Events related with the treatment | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years.
  Adverse events associated with the treatment (s)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Castillo, Dr, Study Director — Scandinavia Pharma
Locations (1):
- Scandinavia Pharma, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No